CLINICAL TRIAL: NCT01555476
Title: Bioequivalence Between an Ibuprofen Suspension and a Reference Formulation. A Study in Healthy Volunteers.
Brief Title: Study to Test the Blood to See if a New Medicine is Likely to Provide Pain Relief Similar to a Product Already Sold in Stores
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IBUPAI1002; 2011-001570-26 (EudraCT Number)
Record Dates: First submitted 2012-03-13; First posted 2012-03-15 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Pain
Keywords: Pharmacokinetics
MeSH Terms: conditions — Pain | interventions — Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A-IBU (Experimental): A single 5 mL dose of 200 mg ibuprofen/5 mL experimental suspension, administered orally, with a 48-hour washout between visits.
  Interventions: Drug: Ibuprofen
- B-IBU (Active Comparator): A single 5 mL dose of 200 mg ibuprofen/5 mL reference suspension, administered orally, with a 48-hour washout between visits
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen — A single 5 mL dose of 200 mg ibuprofen/5 mL experimental suspension, administered orally, with a 48-hour washout between visits
  Other Names: Not yet marketed.
  Arms: A-IBU
Drug: Ibuprofen — A single 5 mL dose of 200 mg ibuprofen/5 mL reference suspension, administered orally, with a 48-hour washout between visits
  Other Names: Nurofen for Children Six Plus
  Arms: B-IBU

SUMMARY:
This study is designed to assess bioequivalence between one test and one reference formulation used for temporary relief of pain. The results will help decide if the new medicine is likely to provide pain relief similar to the product being sold.

DETAILED DESCRIPTION:
The study is a single dose, randomized, two-way crossover study in 32 healthy male and female volunteers, minimum of 14 of each gender. Two doses of study medication will be given as single doses on two separate treatment visits. A washout of at least 48 hours will separate the treatment visits. Each visit will include an overnight fast at the clinic and 19 blood samples drawn for pharmacokinetic analyses. Tolerability of the treatments will be evaluated in terms of reported and observed adverse events (AE).

ELIGIBILITY:
Inclusion Criteria:

* Healthy (per protocol-specified parameters) male or female subjects (14 of each gender) between the ages of 18 and 50 years, inclusive.
* Non- or ex-tobacco user, being defined as someone who completely stopped smoking or using any form of tobacco for at least 12 months before screening visit of this study.
* For females: if not postmenopausal, agrees to use a protocol-specified means of contraception or declared absence of sexual contact with a male partner during the study.
* For males: No pregnant spouse or partner at screening and willingness to protect potential spouse or partner from becoming pregnant during the study.
* Body Mass Index (BMI) within protocol-specified parameters.
* A personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures specified in the protocol.

Exclusion Criteria:

* Evidence or history of an acute or chronic medical or psychiatric condition, laboratory abnormality, or drug use that, in the judgment of the investigator or an authorized physician, may compromise subject safety or the interpretation of results.
* Females: Pregnant or breast-feeding
* Treatment with an investigational drug within 3 months preceding the first dose of study treatment.
* History of regular alcohol consumption outside the protocol-specified allowances.
* Donation or loss of blood within 3 months prior to the first treatment visit if the estimated lost blood volume equaled or exceeded 450 mL.
* Relationship to persons involved directly with the conduct of the study, or their families.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Cmax | During 12 hours post-dose
  Maximum observed plasma concentration (Cmax), is the maximum (peak) concentration (amount of drug) measured in blood plasma after a dose administration.
AUCt | During 12 hours post-dose
  Area under the plasma concentration-vs.-time curve from start of drug administration until last measured concentration (AUCt), is a measure of how much of the drug reaches the bloodstream during the sampling period.

SECONDARY OUTCOMES:
AUC∞ | During 12 hours post-dose
  Area under the plasma concentration-vs.-time curve from start of drug administration and extrapolated to infinity (AUC∞), is a measure of how much of the drug ever reaches the bloodstream.
tmax | During 12 hours post-dose
  The time at which maximum concentration is reached (tmax)
Terminal Elimination Rate Constant (λz) | During 12 hours post-dose
  The terminal elimination rate constant (λz) describes the rate at which a drug is eliminated from the body.
t½ | During 12 hours post-dose
  Terminal half-life (t½) is the time required for the plasma concentration (as well as the amount of drug in the body) to fall by one-half.
Mean Residence Time (MRT) | During 12 hours post-dose
  Mean residence time (MRT) is the mean time a drug molecule resides in the body.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Kruse, PhD, Study Director — McNeil AB
Locations (1):
- McNeil AB Clinical Pharmacology R&D, Lund, Sweden